CLINICAL TRIAL: NCT06102616
Title: Osteocalcin Level in Gingival Clavicular Fluid During Canine Retraction in Periodontal Compromised Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Mohsena Ahmad, Lecturer of Orthodontics, Faculty of Dental Medicine for Girls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12245
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Periodontal Diseases
Keywords: osteocalsin; periodontal compromised teeth; canine retraction
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- periodontal compromised orthodontic pateints (Experimental): periodontal compromised adults female patients with sever dental crowding and seeking for orthodontic treatment
  Interventions: Diagnostic Test: measure Osteocalcin level

INTERVENTIONS:
Diagnostic Test: measure Osteocalcin level — in gingival crevicular fluid before and during orthodontic tooth movement

SUMMARY:
Osteocalcin levels can be measured Gingival crevicular fluid (GCF). Changes in osteocalcin levels can provide important information about the status of bone metabolism and bone remodeling. The levels of this markers in GCF can provide information about the status of bone remodeling in the surrounding bone tissue in periodontal affected teeth.

DETAILED DESCRIPTION:
Osteocalcin levels can be measured using a blood test or by analyzing the levels of osteocalcin in urine or saliva. Changes in osteocalcin levels can provide important information about the status of bone metabolism and bone remodeling. Osteocalcin has been found to be present in Gingival crevicular fluid (GCF), along with other bone metabolism markers such as alkaline phosphatase and tartrate-resistant acid phosphatase. The levels of these markers in GCF can provide information about the status of bone remodeling in the surrounding bone tissue. Orthodontic tooth movement is influenced by the remodelling ability of surrounding bone and soft tissue, such as PDL and gingiva. Bone remodelling occurs in coordination, requiring coupling of bone formation after resorption. Orthodontic force induces an aseptic inflammatory response, involving cytokines and chemokines. . Increased levels of osteocalcin in body fluids indicate abnormal bone turnover activity.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients who were seeking for orthodontic treatment with controlled previous chronic periodontitis.
* Pocket depth of more than 5 mm before receiving non-surgical periodontal treatment or/and Pocket depth of less than 4 mm after periodontal therapy.
* Sever to very sever irregularity of mandibular anterior arch according to Little's irregularity index ranging from 7 to 10 mm with acceptable oral hygiene.
* all the permanent dentition excluding third molars should be present.
* No systemic disease or history of prolonged use of medication interfering with tooth movement as corticosteroids.

Exclusion Criteria:

* Previous orthodontic treatment.
* Patients with aggressive periodontitis or Any smoking habits.
* Pregnant or lactating female patients were excluded.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Osteocalcin levels in gingival crevicular fluid before and during orthodontic tooth movement | at baseline, then after 3 months and after 6 month
  ELISA test to measure osteocalcin in GCF

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dental medicine Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No